CLINICAL TRIAL: NCT04965714
Title: A Pre-Operative Study Evaluating Nivolumab Plus ADI-PEG 20 in Patients With Resectable Hepatocellular Carcinoma
Brief Title: Nivolumab and ADI-PEG 20 Before Surgery for the Treatment of Resectable Liver Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: 0 patient accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-1198; NCI-2021-06214 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-1198 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-07-01; First posted 2021-07-16 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Resectable Hepatocellular Carcinoma
MeSH Terms: interventions — Nivolumab; ADI PEG20

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (nivolumab, pegargiminase) (Experimental): Patients receive nivolumab IV over 30 minutes on day 1 and pegargiminase IM at 2 days before day 1 of cycle 1, day 8 of cycle 1, days 1 and 8 of cycle 2, and day 1 of cycle 3. Treatments repeat every 2 weeks for up to 3 cycles in the absence of disease progression or unacceptable toxicity. Patients then undergo standard of care surgical resection at week 7. A cycle is 14 days.
  Interventions: Biological: Nivolumab; Biological: Pegargiminase; Procedure: Resection

INTERVENTIONS:
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; CMAB819; MDX-1106; NIVO; Nivolumab Biosimilar CMAB819; ONO-4538; Opdivo
Biological: Pegargiminase — Given IM
  Other Names: ADI-PEG 20; pegylated arginine deiminase
Procedure: Resection — Undergo surgical resection
  Other Names: Surgical Resection

SUMMARY:
This phase II trial studies the effect of nivolumab and ADI-PEG 20 before surgery in treating patients with liver cancer that can be removed by surgery (resectable). Immunotherapy with monoclonal antibodies, such as nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. ADI-PEG 20 may stop the growth of tumor cells by blocking some of the proteins needed for cell growth. Giving nivolumab and ADI-PEG 20 before surgery may help control liver cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the safety and tolerability of therapy and assess the pathologic response rate including pathologic complete response (pCR) and degree of necrosis (> 50% in tumor volume) with nivolumab + pegargiminase (ADI-PEG 20) in resectable hepatocellular carcinoma (HCC) in the context of presurgical therapy.

SECONDARY OBJECTIVE:

I. To assess the efficacy of presurgical nivolumab + ADI-PEG 20 therapy in HCC by estimating the time-to-progression (TTP), recurrence-free survival (RFS), and overall survival (OS).

EXPLORATORY OBJECTIVES:

I. To assess the immunological/biomarker changes (pre- versus [vs] post-treatment) in tumor tissues and peripheral blood in response to nivolumab + ADI-PEG 20 in HCC therapy.

II. To explore any potential association between these biomarker measures and antitumor response and immune-related response criteria (irRC) assessed by MD Anderson Department of Diagnostic Imaging.

OUTLINE:

Patients receive nivolumab intravenously (IV) over 30 minutes on day 1 and pegargiminase intramuscularly (IM) at 2 days before day 1 of cycle 1, day 8 of cycle 1, days 1 and 8 of cycle 2, and day 1 of cycle 3. Treatments repeat every 2 weeks for up to 3 cycles in the absence of disease progression or unacceptable toxicity. Patients then undergo standard of care surgical resection at week 7.

After completion of study treatment, patients are followed up at 30 days, then every 12 weeks for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Must give written informed consent prior to initiation of therapy, in keeping with the policies of the institution. Patients with a history of major psychiatric illness must be judged able to fully understand the investigational nature of the study and the risks associated with the therapy
* Must have histologically confirmed HCC (documentation of original biopsy for diagnosis is acceptable if tumor tissue is unavailable) or clinical diagnosis by AASLD (American Association for the Study for Liver Diseases) criteria in cirrhotic subjects (presence of non-rim arterial phase hyperenhancement relative to the liver parenchyma with venous washout for tumors >= 1 cm). For subjects without cirrhosis, histological confirmation is mandatory. The determination of cirrhosis status will ultimately lie in the clinical judgment of the surgical oncologist and medical oncologist involved in the care of the patient
* Must be eligible for liver resection with curative intent; diagnosis must be confirmed by pathologist review of screening biopsy and the determination of resectability status will ultimately lie in the clinical judgment of the surgical oncologist and medical oncologist involved in the care of the patient
* Must have measurable disease defined as a lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) and measures >= 15 mm with conventional techniques or >= 10 mm with more sensitive techniques such as magnetic resonance imaging (MRI) or spiral computed tomography (CT) scan
* Allowed are prior treatments for HCC including prior surgery, radiation therapy, local-regional therapy (ablation or arterial directed therapies), or systemic therapy including sorafenib or chemotherapy. (Prior anti-PD-1 or ADI-PEG 20 therapies are not allowed)
* Must have Eastern Cooperative Oncology Group performance status (ECOG PS) score =< 1
* Absolute neutrophil count >= 1,500/uL (within 14 days of the first dose of study drug)
* Platelets >= 100,000/uL (within 14 days of the first dose of study drug)
* Hemoglobin > 9.0 g/dL (may be transfused or receive epoetin alfa [e.g., Epogen] to maintain or exceed this level) (within 14 days of the first dose of study drug)
* Total bilirubin =< 1.5 mg/dL (within 14 days of the first dose of study drug)
* Serum creatinine =< 1.5 times the upper limit of normal (ULN) or estimated creatinine clearance > 40mL/min (within 14 days of the first dose of study drug)
* Aspartate transaminase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and/or alanine transaminase (ALT) ) (serum glutamate pyruvate transaminase [SGPT]) =< 5 x institutional ULN (within 14 days of the first dose of study drug)
* Serum uric acid =< 10 mg/dL (595 umol/L) (with or without medication control) (within 14 days of the first dose of study drug)
* Must be >= 18 years of age
* Must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) within 24 hours prior to the start of study drug and every 4 weeks while taking nivolumab (for women of childbearing potential [WOCBP])
* Must not be breastfeeding
* Must agree (WOCBP) to follow instructions for method(s) of contraception from the time of enrollment for the duration of treatment with study drug (s) for a total of 12 months post treatment completion. Men who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug(s) plus 5 half-lives of study drug (s) plus 90 days (duration of sperm turnover) for a total of 7 months post-treatment completion

  * NOTE: Azoospermic males and WOCBP who are continuously not heterosexually active are exempt from contraceptive requirements. However, WOCBP must still undergo pregnancy testing as described in these sections. Investigators shall counsel WOCBP and male subjects who are sexually active with WOCBP on the importance of pregnancy prevention and the implications of an unexpected pregnancy Investigators shall advise WOCBP and male subjects who are sexually active with WOCBP on the use of highly effective methods of contraception. Highly effective methods of contraception have a failure rate of < 1% per year when used consistently and correctly. At a minimum, subjects must agree to the use of two methods of contraception, with one method being highly effective and the other method being either highly effective or less effective as listed below:

HIGHLY EFFECTIVE METHODS OF CONTRACEPTION

* Male condoms with spermicide
* Hormonal methods of contraception including combined oral contraceptive pills, vaginal ring, injectables, implants, and intrauterine devices (IUDs) such as Mirena by WOCBP subject or male subject's WOCBP partner.
* Nonhormonal IUDs, such as ParaGard
* Tubal ligation
* Vasectomy
* Complete Abstinence*
* Complete abstinence is defined as complete avoidance of heterosexual intercourse and is an acceptable form of contraception for all study drugs. Abstinence is only acceptable when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (eg, calendar, ovulation, symptothermal, profession of abstinence for entry into a clinical trial, post-ovulation methods) and withdrawal are not acceptable methods of contraception. Subjects who choose complete abstinence are not required to use a second method of contraception, but female subjects must continue to have pregnancy tests. Acceptable alternate methods of highly effective contraception must be discussed in the event that the subject chooses to forego complete abstinence.

LESS EFFECTIVE METHODS OF CONTRACEPTION

* Diaphragm with spermicide
* Cervical cap with spermicide
* Vaginal sponge
* Male condom without spermicide*
* Progestin only pills by WOCBP subject or male subject's WOCBP partner
* Female condom*
* A male and female condom must not be used together

  * Must not have received prior anticancer therapy with ADI-PEG 20 or anti-PD1 for HCC. Must not be receiving any concomitant systemic therapy for HCC

Exclusion Criteria:

* Has any other malignancy from which the patient has been disease-free for less than 2 years (exceptions: non-melanoma skin cancer or in situ carcinoma of any site are allowed)
* Has an organ allograft(s)
* Has had a major surgical procedure, open biopsy, or significant traumatic injury with poorly healed wound within 6 weeks prior to first dose of study drug; or anticipates needing for a major surgical procedure during the course of the study (other than defined by protocol such as the pre-treatment fine needle aspirations or core biopsies) within 7 days prior to first dose of study drug
* Has a history of inflammatory bowel disease (including Crohn's disease and ulcerative colitis) or a history of autoimmune disease (e.g., rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, autoimmune vasculitis [e.g., Wegener's granulomatosis])
* Has a history of testing positive for human immunodeficiency virus or has acquired immunodeficiency syndrome (AIDS)
* Has any underlying medical condition, which in the opinion of the investigator, will make the administration of study drug hazardous or will obscure the interpretation of adverse events, such as a condition associated with frequent diarrhea
* Has a known risk factor for bowel perforation including a history of acute diverticulitis, abdominal fistula, gastrointestinal perforation, intra-abdominal abscess, or gastrointestinal obstruction
* Has a primary brain tumor (excluding meningiomas and other benign lesions), any brain metastases, leptomeningeal disease, seizure disorders not controlled with standard medical therapy, or (within the past year) a history of stroke
* Has a history of serious systemic disease, including myocardial infarction or unstable angina within the last 12 months; a history of hypertensive crisis or hypertensive encephalopathy, uncontrolled hypertension (blood pressure of > 140/90 mmHg) at the time of enrollment; New York Heart Association (NYHA) grade II or greater congestive heart failure, unstable symptomatic arrhythmia requiring medication (patients with chronic atrial arrhythmia, i.e., atrial fibrillation or paroxysmal supraventricular tachycardia are eligible); significant vascular disease or symptomatic peripheral vascular disease
* Has a history of other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that might affect the interpretation of the results of the study or render the subject at high risk from treatment complications
* Is receiving a high dose steroid (e.g., > 10 mg prednisone daily or equivalent) or other more potent immune suppression medications (e.g., infliximab)
* Has had influenza-, hepatitis-, or other vaccines within a month prior to initiation of study drugs
* Has had a clinical history of coagulopathy, bleeding diathesis or thrombosis within the past year
* Has a serious, non-healing wound, ulcer, or bone fracture
* Is pregnant (positive pregnancy test) or lactating
* Had a prior orthotropic liver transplantation
* Has cirrhosis and severe synthetic liver dysfunction (Child Pugh B-C)
* Has received any complementary medications (e.g., herbal supplements or traditional Chinese medicines) intended to treat the disease under study unless patients agree to stop the complementary medicines at least 14 days before the first study dose. Such medications are permitted if they are used as supportive care
* Has received any live / attenuated vaccine (e.g., varicella; zoster; yellow fever; rotavirus; oral polio; or and measles, mumps, rubella) within a month prior to initiation of study drug or during treatment are excluded
* Must not be scheduled to receive another experimental drug while on this study
* Must not require ongoing anticoagulation therapy (although aspirin and pre- and postsurgical prophylactic anti coagulation treatment are permitted
* Must not require total parenteral nutrition
* Not able to be compliant with the appointments required in this protocol
* Has a history of seizure disorder not related to underlying cancer
* Has a known allergy to pegylated compounds
* Has a known allergy to E. coli drug products (such as granulocyte-macrophage colony stimulating factor)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-04-13 (Actual); Primary Completion 2023-02-10 (Actual); Study Completion 2023-02-10 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 30 days post-treatment
  Safety will be recorded through the incidence of AEs, serious (S)AEs and specific laboratory abnormalities (worst grade). Toxicities will be graded using the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. Will tabulate AEs with frequency and percentage and will summarize them by severity and their relations to the study treatments, and will estimate the success rate along with the 95% exact confidence interval.
Rate of pathologic complete response | Up to 2 years post-treatment
  Pathological response rate will be estimated along with the 95% confidence interval (95% CI).
Necrosis of tumors | Up to 2 years post-treatment

SECONDARY OUTCOMES:
Time-to-progression (TTP) | Up to 2 years post-treatment
  TTP is defined as the time from the start of study drug to the first documented tumor progression or recurrence of tumor as determined by the investigator using Response Evaluation Criteria in Solid Tumors 1.1 or Immune-Related Response Criteria (irRC) criteria. Will be estimated by the Kaplan-Meier method.
Recurrent-free survival (RFS) | From surgery to date of a recurrent disease or date of death whichever occurs first if patients have an event, or to the last follow-up date if patients are alive without RD, assessed up to 2 years
  RFS will be estimated by the Kaplan-Meier method.
Overall survival (OS) | From the initiation of the study combination to the date of death, assessed up to 2 years
  OS will be estimated by the Kaplan-Meier method.

OTHER OUTCOMES:
Immune biomarker analysis | Up to 2 years post-treatment
  Will use descriptive statistics to summarize expressions of markers at each time point and will use paired t-test or Wilcoxon signed rank test to evaluate the pre- and post- treatment changes in immune biomarkers, including CD8+/Treg ratio. To correlate markers with response, will fit logistic regression models or use a Fisher's exact test. For longitudinal measurements, we will use logistic regression models including random effects to account for within-patient correlation. To evaluate marker changes over time, will fit linear mixed models with random effects to account for within-patient correlation.

CONTACTS AND LOCATIONS:
Overall Officials: Sunyoung Lee, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org